CLINICAL TRIAL: NCT02522754
Title: Study to Determine if Intranasal Proteosome-Adjuvanted Trivalent Influenza Vaccine is Safe, Immunogenic and Efficacious in the Influenza Human Viral Challenge Model
Brief Title: Development of an Intranasal Proteosome Influenza Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hvivo (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, R Lambkin-Williams, Chief Scientist, Hvivo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IDB 004 IDB 005
Record Dates: First submitted 2015-07-28; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo Protesomal Vaccine
- Protesomal Vaccine 1 x 30 µg (Experimental): Protesomal Vaccine 1 x 30 µg
  Interventions: Biological: Experimental: Protesomal Vaccine 1 x 30 µg
- Protesomal Vaccine 2 x 30 µg (Experimental): Protesomal Vaccine 2 x 30 µg
  Interventions: Biological: Experimental: Protesomal Vaccine 2 x 30 µg
- Protesomal Vaccine 2 x 15 µg (Experimental): Protesomal Vaccine 2 x 15 µg
  Interventions: Biological: Experimental: Protesomal Vaccine 2 x 15 µg

INTERVENTIONS:
Biological: Placebo Protesomal Vaccine — Intranasal vaccine Protesomal Vaccine
  Other Names: Placebo
  Arms: Placebo
Biological: Experimental: Protesomal Vaccine 1 x 30 µg — Experimental: Protesomal Vaccine 1 x 30 µg
  Arms: Protesomal Vaccine 1 x 30 µg
Biological: Experimental: Protesomal Vaccine 2 x 30 µg — Experimental: Protesomal Vaccine 2 x 30 µg
  Arms: Protesomal Vaccine 2 x 30 µg
Biological: Experimental: Protesomal Vaccine 2 x 15 µg — Experimental: Protesomal Vaccine 2 x 15 µg
  Arms: Protesomal Vaccine 2 x 15 µg

SUMMARY:
A study to compare multiple dosage regimes of a protesomal intranasal vaccine.

DETAILED DESCRIPTION:
A Proteosome-adjuvanted trivalent inactivated influenza vaccine (P-TIV) administered intra-nasally was shown to be effective, safe, well tolerated, immunogenic - in both systemic and mucosal compartments - and effective at preventing influenza illness.

In two separate studies using the Human Viral Challenge Model, subjects were selected for susceptibility to A/Panama/2007/1999 (H3N2) virus and then dosed with one of three regimens: (A/New Caledonia/20/1999 (H1N1), A/Panama/2007/1999 (H3N2), B/Victoria/504/2000 or B/Shangdong/7/1997) or placebo via a nasal spray. One or two doses were given, 14 days apart, before subjects were challenged with ~8.5 x 105 EID¬50 of A/Panama/2007/1999 (H3N2) virus. Immune responses to the vaccine antigens were measured, namely serum IgG (via the aemagglutination inhibition assay (HAI)) and nasal wash secretory IgA (sIgA) antibodies (via ELISA). Viral titres in nasal washes and symptoms of influenza illness were assessed after viral challenge and compared.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy adults as determined by medical history, physical examination, serology (HIV and Hepatitis B and C) and clinical laboratory tests.
* Female subjects were required to provide of a history of reliable contraceptive practice.
* Susceptibility to A/Panama/2007/1999 (H3N2) (a serum reciprocal HAI titre ≤10) was confirmed at screening. -

Exclusion Criteria:included;

* asthma,
* hypersensitivity to mercurials or chicken eggs,
* anatomic or neurologic abnormality impairing the gag reflex or contributing to aspiration, * chronic nasopharyngeal complaints,
* abnormal electrocardiogram (ECG),
* febrile illness or significant symptoms of upper respiratory infection on the day of vaccination or between admission to quarantine and administration of the challenge inoculum.
* Subjects using medication or other products for rhinitis or nasal congestion,
* Subject who had received systemic glucocorticoids within 1 month, or cytotoxic or immunosuppressive drugs within 6 months of the study start.
* Subjects agreed not to smoke during the quarantine phase.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2002-01; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Reduction in Influenza Like Illness in those with laboratory confirmed influenza | Within the duration of infection, approx 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Rob Lambkin-Williams, PhD, Principal Investigator — PI

REFERENCES:
- [Derived] Lambkin-Williams R, Gelder C, Broughton R, Mallett CP, Gilbert AS, Mann A, He D, Oxford JS, Burt D. An Intranasal Proteosome-Adjuvanted Trivalent Influenza Vaccine Is Safe, Immunogenic & Efficacious in the Human Viral Influenza Challenge Model. Serum IgG & Mucosal IgA Are Important Correlates of Protection against Illness Associated with Infection. PLoS One. 2016 Dec 22;11(12):e0163089. doi: 10.1371/journal.pone.0163089. eCollection 2016. PMID 28005959